CLINICAL TRIAL: NCT03844997
Title: Phase I/II Trial of CPX-351 + Palbociclib in Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sudipto Mukherjee, MD, PhD, MPH (Other)
Responsible Party: Sponsor-Investigator, Sudipto Mukherjee, MD, PhD, MPH, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CASE1918
Record Dates: First submitted 2019-01-28; First posted 2019-02-19 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — palbociclib; CPX-351

STUDY DESIGN:
Intervention Model Description: This is a single arm, open label study of the combination of Palbociclib with CPX-351 in adults with AML. The trial consists of two components: phase I to evaluate the safety with dose escalation of Palbociclib in combination with CPX-351 and phase II to evaluate the overall response rate of the combination in the targeted patient population. A cycle is 28 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Palbociclib + CPX-351 (Experimental): Palbociclib will be administered orally on day -1 and -2 at 125 mg PO during the phase IIaportion (dose level 0).Day 0 will be rest and then CPX-351 at 100 u/m2 will be started on days 1, 3, and 5 along with Palbociclib day 2, 4, and 6 followed by rest/monitoring period (day 7-28).
  If Grade 3-4 non-hematologic toxicity is observed in 1 or less of 6 patients treated, the study will move to Phase IIb. If Grade 3-4 non-hematologic toxicity is observed in 2 or more of 6 patients treated, 6 additional patients will be treated on the Phase IIa portion at a lower dose level (100 mg po) until a Phase IIb safe dose schedule is defined at which 1 or less out of 6 patients on the Phase IIa experience Grade 3-4 non-hematologic toxicity. After the Phase IIa portion ensures safety, the study will proceed with phase IIb. The phase IIb component is a Simon 2-stage design trial whose objective is to assess the clinical efficacy of the combination of Palbociclib and CPX-351.
  Interventions: Drug: Palcociclib; Drug: CPX-351

INTERVENTIONS:
Drug: Palcociclib — Palbociclib is an investigational (experimental) drug that works to induce early G1 arrest by inhibiting CDK4/6, which are two types of CDKs that are overexpressed in AML cell cancer lines. Palbociclib is experimental because it is not approved by the Food and Drug Administration (FDA).
  Palbociclib will be supplied as capsules or tablets containing 125 mg equivalents of Palbociclib free base
  Other Names: IBRANCE
Drug: CPX-351 — CPX-351 (daunorubicin and cytarabine) liposome for injection is a combination of daunorubicin and cytarabine in a 1:5 molar ratio encapsulated in liposomes for intravenous administration. CPX-351 is an investigational (experimental) drug that works as formulation of a fixed combination of the antineoplastic drugs cytarabine and daunorubicin. CPX-351 is experimental because it is not approved by the Food and Drug Administration (FDA).
  Other Names: VYXEOS

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Palbociclib in combination with investigational (experimental) drug, CPX-351 and evaluate the efficacy of Palbociclib in combination with chemotherapy as measured by overall response rate (ORR), i.e. complete response (CR) and CR with incomplete blood count recovery (CRi) by 2003 IWG criteria.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the safety and tolerability of Palbociclibin combination with CPX-351, and to evaluate the efficacy of Palbociclibin combination with chemotherapy as measured by overall response rate (ORR), i.e. complete response (CR) and CR with incomplete blood count recovery (CRi) by IWG criteria.

CPX-351 is an investigational drug that works as formulation of a fixed combination of the antineoplastic (acting to prevent, inhibit or halt the development of a neoplasm (a tumor)) drugs cytarabine and daunorubicin.

Palbociclibis an investigational drug that works to induce early G1 arrest by inhibiting CDK4/6, which are two types of CDKs that are overexpressed in AML cell cancer lines.

CPX-351 and Palbociclib is experimental because it is not approved by the Food and Drug Administration (FDA).

This is a single arm, open label study of the combination of Palbociclib with CPX-351 in adults with AML. The trial consists of two components: phase I to evaluate the safety with dose escalation of Palbociclib in combination with CPX-351 and phase II to evaluate the overall response rate of the combination in the targeted participant population.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed acute myeloid leukemia according to 2016 WHO criteria(excluding APL [AML-M3]).
* Eastern Cooperative Oncology Group (ECOG) Performance Status <2
* Subjects must have normal organ function as defined below:
* Total bilirubin <2 times upper limit of normal ((≤ 3 x ULN if considered to be due to leukemic involvement or Gilbert's syndrome) or if higher than 2 times upper limit of normal with approval from the PI
* Serum Creatinine <2 x ULNor if higher than 2 times upper limit of normal with approval from the PI
* Left ventricular ejection fraction of ≥45%
* Patients with secondary AML arising out of MDS (all subtypes under WHO classification), chronic myelomonocytic leukemia (CMML) and therapy-related AML are eligible.
* Women of childbearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment. All men and women of childbearing potential must use acceptable methods of birth control throughout the study
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment with CPX-351, Palbociclib or other cell cycle inhibitors.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that, in the view of the treating physician, would place the participant at an unacceptable risk if he or she were to participate in the study or would prevent that person from giving informed consent.
* Any active malignancy (unrelated, non-hematological malignancy) diagnosed within the past 6 months of starting the study drug (other than curatively treated carcinoma-in-situ of the cervix or non-melanoma skin cancer).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CPX-351, Palbociclib or other cell cycle inhibitors.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known history of HIV or active hepatitis B or C.
* No major surgery within 2 weeks prior to study enrollment.
* Pregnancy or breast feeding
* Male and female patients who are fertile who do not agree to use an effective barrier methods of birth control (i.e. abstinence) to avoid pregnancy while receiving study treatment.
* Acute promyelocytic leukemia (APL)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudipto Mukherjee, MD, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Palbociclib was given at dose level 1 (75 mg po) on day -1 and -2, day 0 was rest and then CPX-351 (daunorubicin 44 mg/m2 and cytarabine 100 mg/m2) was started on day 1, 3, and 5 along with Palbociclib on day 2, 4, and 6 followed by rest/monitoring period (days 7-35)
- Phase II: Patients received 1-2 induction courses of the combination of Palbociclib and 125mg of CPX-351.
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 9 | 26
Completed | 9 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Palbociclib will be given at dose level 1 (75 mg po) on day -1 and -2, day 0 will be rest and then CPX-351 (daunorubicin 44 mg/m2 and cytarabine 100 mg/m2) will be started on day 1, 3, and 5 along with Palbociclib on day 2, 4, and 6 followed by rest/monitoring period (days 7-35)
- Phase II: Patients will receive 1-2 induction courses of the combination of Palbociclib and CPX-351.
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 9 | 26 | 35
Age, Customized [Median (Full Range); unit: years] | 47 [30 to 68] | 56 [27 to 65] | 56 [27 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 14 | 18
  Male | 5 | 12 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 9 | 24 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 7 | 22 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
History of Cancer [Count of Participants; unit: Participants]
  No cancer | 5 | 3 | 8
  AML | 2 | 22 | 24
  MDS | 0 | 1 | 1
  MPN | 1 | 0 | 1
  Other cancer | 1 | 0 | 1
AML(Acute Myeloid Leukemia) Classification [Count of Participants; unit: Participants]
  Unknown | 2 | 0 | 2
  AML not otherwise specified | 3 | 16 | 19
  AML with certain genetic abnormalities | 2 | 8 | 10
  AML with myelodysplasia-related changes | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Experimental Dose of Palbociclibin Combination With CPX-351 as Measured by Number of Participants With Dose Limiting Toxicities.
Description: If Grade 3-4 non-hematologic toxicity is observed in 1 or less of 6 patients treated, the dose of the study drug will be considered safe/tolerable. If Grade 3-4 non-hematologic toxicity is observed in 2 or more of 6 patients treated, 6 additional patients will be treated on the Phase IIa portion at a lower dose level (100 mg po).
Time Frame: Between days 28-35 of starting treatment
Population: Safety and tolerability only measured for Phase I
Measure: Count of Participants; unit: Participants
Groups:
- Phase II: Participants received 1-2 induction courses of the combination of Palbociclib and CPX-351
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 9 | 0
Participants | 0 |

2. Primary Outcome: Efficacy of Palbociclibin Combination With Chemotherapy as Measured by Overall Response Rate (ORR).
Description: Efficacy of Palbociclibin combination with chemotherapy as measured by overall response rate (ORR) which is defined as complete response (CR) and CR with incomplete blood count recovery (CRi) by IWG criteria.
  Complete remission is defined as: Bone marrow blasts <5%; absence ofcirculating blasts and blasts with Auerrods; absence of extramedullarydisease; absolute neutrophil count >1.0x 109/L (1,000/μL); platelet count >100 x109/L (100,000/μL)
  and
  CR with incomplete blood count recovery is defined as: All CR criteria except for residualneutropenia [<1.0 x 109/L (1,000/μL)] orthrombocytopenia [<100 x 109/L(100,000/μL)].
  Either of these responses will constitute ORR.
Time Frame: Up to 2 years from end of treatment, up to 27 months
Population: ORR was measured only for Phase II
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 0 | 26
Participants |  | 22

3. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as the time it takes from the start date of the treatment to the date of achievement of response (as per the definition of response mentioned in the 2003 IWG criteria).
Time Frame: Up to 2 years from end of treatment
Measure: Geometric Mean (Full Range); unit: Days
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 6 | 22
Days | 43.37 [35 to 62] | 41.27 [33 to 103]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is measured between the date of response to date of loss of response.
Time Frame: Up to 2 years from end of treatment
Measure: Geometric Mean (Full Range); unit: Days
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 6 | 22
Days | 302.91 [119 to 720] | 523.7 [66 to 735]

5. Secondary Outcome: Event-free Survival (EFS)
Description: EFS measured from the date of entry into a study to the date of primary refractory disease, or relapse from CR, or CRi, or death from any cause; patients not known to have any of these events are censored on the date they were last examined
Time Frame: Up to 2 years from end of treatment
Measure: Geometric Mean (Full Range); unit: Days
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 9 | 26
Days | 188.23 [20 to 767] | 406.09 [42 to 787]

6. Secondary Outcome: Overall Survival (OS) Probability
Description: OS probability measured from the date of entry into a clinical trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive
Time Frame: Up to 2 years from end of treatment, up to 27 months
Measure: Number; unit: percentage of paticipants
Groups:
- Phase II: Patients received 1-2 induction courses of the combination of Palbociclib and CPX-351.
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 9 | 26
percentage of paticipants | 25 | 76

ADVERSE EVENTS:
Time Frame: All adverse events were collected through 30 days after the final dose of study drug, up to 100 days, all cause mortality was assessed through 2 years from end of treatment
Groups:
- Phase I: Palbociclib was administered orally on day -1 and -2 at 125 mg PO during the phase IIaportion (dose level 0).Day 0 will be rest and then CPX-351 at 100 u/m2 will be started on days 1, 3, and 5 along with Palbociclib day 2, 4, and 6 followed by rest/monitoring period (day 7-28).
Arm/Group | Phase I | Phase II
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/9 | 3/26
Other Adverse Events (participants affected / at risk) | 9/9 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=9) | Phase II (N=26)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=9) | Phase II (N=26)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (5) | 16 (42)
Alkaline phosphatase increased (Investigations) | 5 (7) | 9 (17)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 9 (66) | 20 (47)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Anxiety (Psychiatric disorders) | 2 (4) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (6) | 16 (43)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (12)
Bacteremia (Infections and infestations) | 1 (1) | 4 (4)
Belching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (6) | 8 (14)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (3)
Cardiac troponin T increased (Investigations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Chest wall pain (Cardiac disorders) | 0 (0) | 1 (2)
Chills (General disorders) | 2 (2) | 7 (9)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6) | 12 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 11 (15)
Creatinine increased (Investigations) | 4 (4) | 8 (16)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 12 (14)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 8 (8)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 3 (5)
Edema face (General disorders) | 0 (0) | 2 (2)
Edema limbs (Musculoskeletal and connective tissue disorders) | 3 (3) | 11 (11)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 12 (14)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 12 (13)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 24 (36)
Fever (General disorders) | 4 (10) | 4 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2)
Floaters (Eye disorders) | 0 (0) | 4 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 2 (2)
Generalized edema (General disorders) | 0 (0) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Genital edema (General disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (7) | 14 (19)
Hematoma (Vascular disorders) | 0 (0) | 2 (3)
Hematuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 5 (12)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (12) | 12 (17)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 7 (9) | 18 (33)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 6 (8) | 14 (28)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 14 (26)
Hypotension (Vascular disorders) | 2 (3) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 5 (8)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Infusion site extravasation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 7 (7)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 1 (1) | 4 (4)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (5)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2) | 5 (8)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 11 (14)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (7) | 15 (20)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 8 (19) | 13 (30)
Non-cardiac chest pain (General disorders) | 0 (0) | 8 (12)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Oral pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Otitis media (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 2 (2) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1) | 2 (2)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 8 (38) | 23 (79)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (11)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (6) | 21 (34)
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Salivary gland infection (Infections and infestations) | 0 (0) | 1 (1)
Scleral disorder (Eye disorders) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus tachycardia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (4) | 10 (12)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Vascular disorders) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 1 (2)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (4)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 9 (25) | 21 (67)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT03844997/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT03844997/ICF_001.pdf